CLINICAL TRIAL: NCT02567110
Title: Inflammation-Induced Central Nervous System (CNS) Glutamate as a Function of Depression in Middle Age
Brief Title: Magnetic Resonance Spectroscopy (MRS) in Midlife Depression
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ebrahim Haroon, Associate Professor, Emory University
Other Study IDs: IRB00083464; 5R01MH107033-04 (NIH)
Record Dates: First submitted 2015-09-29; First posted 2015-10-02 (Estimated); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Depression; Depression Bipolar
Keywords: Mid-life Depression; Bipolar Disorder; DSM-5 MDE; Inflammation; CNS Glutamate
MeSH Terms: conditions — Depression; Bipolar Disorder; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — inflammatory gene expression studies, APOE4 genotyping
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with Major Depression: Participants with major depression will complete neurocognitive and psychiatric assessments, complete self-report forms and undergo Magnetic Resonance Imaging scans. Blood and spinal fluid specimens will also be collected for estimation of inflammatory markers.
- Participants without Depression: Participants without depression will complete neurocognitive and psychiatric assessments, complete self-report forms and undergo Magnetic Resonance Imaging scans. Blood and spinal fluid specimens will also be collected for estimation of inflammatory markers.

SUMMARY:
The purpose of this study is to determine the impact of inflammation on central nervous system (CNS) glutamate, white matter pathology and alterations in behavior and cognition in middle-aged patients with major depression. Depression is associated with significant alterations in glutamate concentrations and white matter integrity, which has been associated with decreased antidepressant response, poor functional outcome, and cognitive impairment.

DETAILED DESCRIPTION:
This study involves behavioral assessments, neurocognitive testing, blood sampling and magnetic resonance imaging (MRI) scanning. Goals of this study are to determine the impact of inflammation on glutamate concentrations in the basal ganglia and on the integrity of white matter tracts in the basal ganglia and other subcortical regions of middle-aged depressed versus non-depressed individuals and to associated the impact of glutamate and white matter changes on behavioral symptoms among the same group of patients.

ELIGIBILITY:
Inclusion Criteria for Participants with Depression:

* Willing and able to give written informed consent
* Meet criteria for Major Depression per DSM-V criteria using Structured Clinical Interview for DSM-V (SCID-V) and a score ≧18 on the 17-item Hamilton Rating Scale for Depression (HAMD).
* Absence of significant suicidal ideation, determined by the Columbia Suicide Severity Rating Scale - Screen Version (CSSRS)
* Meets MRI scanning safety requirements:

  * Absence of embedded MR-unsafe metallic objects
  * Location and quantity of MR-safe metallic objects will minimally impact rigor/reproducibility standards of the MR data (as determined by the PI in consultation with the neuroimaging team)

Specific Inclusion Criteria for Controls:

* Criteria for major depression not met per the SCID-V
* HAMD scores ≦7
* Absence of any Axis I pathology

Exclusion Criteria:

* Unstable cardiovascular, endocrinologic, hematologic, hepatic, renal, or neurologic disease as evidenced by any of the following:

  * Clinically significant abnormalities in lab values, medical history and physical exam as determined by PI or their designee
  * Changes in medications prescribed for chronic medical illnesses within past 4 weeks,
  * Hospitalization or drastic medical changes within past 4 weeks
* Cognitive impairment as defined by:

  * Score of < 28 on Mini-mental exam (MMSE)
  * Below 8th grade reading ability as defined by Wide Range Achievement Test-3 (WRAT3) score
* Presence of psychosis (lifetime) / mania (current) as defined by:

  * Lifetime diagnosis of psychotic disorders SCID-V
  * SCID-V criteria for current mania/hypomania within the current episode
* Clinically significant substance abuse within the past 6 months as defined by meeting the SCID-V threshold of severity for > 4/11 criteria for substance abuse disorder
* Presence of active symptoms of an eating disorder as defined by:

  * SCID-V diagnosis of Anorexia or bulimia nervosa.
  * Binge eating and/or purging behavior in the absence of mood alterations or precipitating stress (bingeing within the current episode of mood symptoms will not be exclusionary)
* Presence of significant psychiatric comorbidities during current episode:

  * Primary diagnosis of anxiety-spectrum disorders (panic, generalized anxiety, social phobia etc.), PTSD, OCD based on SCID-V criteria
  * Severity of above diagnoses exceeds that of major depression based on assessments by the PI and the Study Team members
* Severe Axis II personality pathology as determined by a clinician
* Use of immune-active medications:

  * Continuous use of prescribed, standard dose non-steroidal anti-inflammatory (NSAIDs) excluding 81 mg of aspirin within past 1 week and PRN use of NSAIDs within past 72 hours
  * Intake of antibiotics within the past 2 weeks
  * Immunization (including seasonal flu) within the past 2 weeks
  * Use of topical or inhaled steroids within 72 hours unless otherwise approved by PI
  * Use of systemic steroids (oral or parenteral) within past 6 months
  * Patients taking herbal supplements with currently known effects on immune system including omega-3 supplements within 2 weeks or probiotics prior to research blood draws and scan unless approved by PI.
* Use of psychotropics:

  * Daily intake of standard doses of antidepressants, mood stabilizers, antipsychotics, psychostimulants within 2 weeks (8 weeks for fluoxetine) prior to initiation of study procedures (scan and research blood sampling)
  * Daily/clinically significant use of sedative-hypnotics and tranquilizers and opiates as determined by PI
  * PRN use of sedative/hypnotics, benzodiazepines exceeding equivalent of clonazepam 1mg within 48 hours of study visit.
* Cancer and autoimmunity:

  * Life time history of diagnosis and/or treatment of cancers other than basal cell carcinoma
  * Life time history of diagnosis and/or treatment of autoimmune disorders including but not restricted to multiple sclerosis, inflammatory bowel disease, systemic lupus erythematosus, rheumatoid arthritis, and Hashimoto's thyroiditis

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female patients who have a diagnosis of depression or bipolar depression and men and women without a diagnosis of depression or bipolar depression in the control group
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2016-07; Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Levels of Glutamate in the basal ganglia | Day 1 (Day after Screening)
  Single-voxel MRS (Magnetic Resonance Spectroscopy) scans will be done to determine the glutamate levels in the basal ganglia. MRS uses a magnetic field to look at magnetic nuclei which absorb and re-emit electromagnetic energy in the presence of the magnetic field. By looking at the peaks in the resultant spectra, the structure and concentrations of metabolite can be determined.

SECONDARY OUTCOMES:
Neurocognitive Testing | Day 1 (Day after Screening)
  The Cambridge Neuropsychological Test Automated Battery (CANTAB) instrument will be used to evaluate multiple cognitive domains including reaction time, attention and information processing. Findings will be compared between depressed participants and healthy controls.
Hamilton Rating Scale for Depression (HAM-D-17) Score | Day 1 (Day after Screening)
  Clinician rated depression will be examined with the Hamilton Rating Scale for Depression (HAM-D-17). The HAM-D-17 is a 17-item scale used to assess present-state depression. Responses are on a 3 or 5-point scale (depending on the item) where 0 = absence of the problem and 3 or 5 = severe problem. Total raw scores range from 0 to 50 where higher scores indicate increased symptoms of depression.
Disease affecting white matter connecting frontal cortex to other regions of the brain | Day 1 (Day after Screening)
  Diffusion tensor imaging (DTI) scans will be obtained to to study white matter disease in frontal cortex.

CONTACTS AND LOCATIONS:
Overall Officials: Ebrahim Haroon, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory Clinic, Atlanta, Georgia
  - Emory University Hospital Clinical Research Network, Atlanta, Georgia
  - Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Undecided